CLINICAL TRIAL: NCT06033820
Title: A Prospective, Single Arm, Open Label Study to Evaluate the Safety and Efficacy of Zanubrutinib, Lenalidomide With R-ICE Chemotherapy for Relapsed/Refractory Diffuse Large B-cell Lymphoma.
Brief Title: Zanubrutinib+Lenalidomide+R-ICE in Relapsed/Refractory DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-0229
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Large B-cell Lymphoma Recurrent; Diffuse Large B Cell Lymphoma Refractory
Keywords: diffuse large B-cell lymphoma; Zanubrutinib; Lenalidomide; Salvage therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZR2-ICE Group (Experimental): All patients will receive 3 cycles of ZR2-ICE immunochemotherapy every three weeks.
  Interventions: Drug: ZR2-ICE

INTERVENTIONS:
Drug: ZR2-ICE — * Drug: zanubrutinib Oral Capsule
  * Drug: lenalidomide Oral Capsule
  * Drug: R-ICE chemotherapy

SUMMARY:
This is a prospective, single center, single arm, open label study of zanubrutinib, lenalidomide in combination with Rituximab-ICE for treatment of relapsed/refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 75 years 2. Histologically confirmed diagnosis of DLBCL, CD20 positive 3. Patients received at least one systemic regimens for the treatment of DLBCL, and one therapy line must have included a CD20-targeted therapy.

4. Relapsed or refractory disease 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. 6. Measurable disease on cross section imaging by PET and/or CT that is at least 1.5 cm in the longest diameter and measurable in two perpendicular dimensions as defined by IWG criteria.

7. Patients must meet the following laboratory criteria at screening, including:

1. Absolute neutrophil count (ANC) ≥1.5 x 109/L or ≥0.75 x 109/L if bone marrow involvement
2. Platelets ≥90 x 109/L or ≥50 x 109/L if bone marrow involvement
3. Hemoglobin ≥75 g/dL or ≥50 g/dL if bone marrow involvement
4. Total bilirubin ≤2.5 x upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of hepatic involvement.
5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤3 x (ULN) or < 5 x ULN if hepatic involvement.
6. Creatinine Clearance Rate ≥60 mL/min.
7. INR ≤1.5 x ULN and aPTT ≤1.5 x ULN 8. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. For females, these restrictions apply for 3 month after the last dose of study drug.

9. Male subject agrees to use an acceptable method for contraception for the duration of the study. Men must agree to not donate sperm during and after the study. For males, these restrictions apply for 3 months after the last dose of study drug.

10. Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, and are willing to participate in the study. Must be able to adhere to study visit schedules and other protocol requirements.

Exclusion Criteria:

1. Patients who have a history of "double/triple hit" genetics. 2. Patients who have, within 14 days prior to Day 1 dosing:

1. not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma specific therapy.
2. undergone major surgery or suffered from significant traumatic injury.
3. received live vaccines.
4. required parenteral antimicrobial therapy for active, intercurrent infections. 3. Patients who have use investigational agents within the period ≤ 3 months prior to Day 1 dosing.

4. Patients who have,

1. Adverse events (AEs) due to previous anti-tumor therapy have not recovered
2. Known allergy or sensitivity to any drug contained in the regimen
3. have undergone ASCT within the period ≤3 months prior to signing the informed consent form.
4. have undergone previous allogenic stem cell transplantation.
5. have a history of deep venous thrombosis/embolism and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period.
6. concurrently use other anticancer or experimental treatments. 5. Coexistent second malignancy or history of prior malignancy within previous 5 years.

6. Patients who have,

1. Known history of active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
2. Known history of human immunodeficiency virus (HIV) infection.
3. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.
4. History of gastrointestinal disorder or defect that would interfere with the absorption of the study drug.
5. Patients with history of severe hemorrhagic disorders.
6. History of stroke or intracranial hemorrhage within 6 months prior to registration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 9 weeks
  To evaluate the efficacy in terms of objective response rate including CR and PR rate after three cycles of ZR2-ICE

SECONDARY OUTCOMES:
Complete remission rate (CR) | 9 weeks
  To evaluate the efficacy in terms of Complete Response Rate after three cycles of ZR2-ICE
DOR | Up to 2 years
  Among participants who experience an objective response, DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression
Progression-free survival | Up to 2 years
  Progression-free survival is defined as the time from enrolment to progression or death due to any cause. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Overall survival | Up to 2 years
  Overall survival is defined as the time from enrolment to death due to any cause.
Safety Management Study | Up to 100 days
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No